CLINICAL TRIAL: NCT03303950
Title: Busulfan, Fludarabine, Donor Stem Cell Transplant, and Cyclophosphamide in Treating Participants With Multiple Myeloma or Myelofibrosis
Brief Title: Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI98381
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Results first posted 2020-05-27 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Anemia; ASXL1 Gene Mutation; EZH2 Gene Mutation; IDH1 Gene Mutation; IDH2 Gene Mutation; Plasma Cell Myeloma; Primary Myelofibrosis; Recurrent Plasma Cell Myeloma; Secondary Myelofibrosis; Thrombocytopenia
MeSH Terms: conditions — Anemia; Multiple Myeloma; Primary Myelofibrosis; Thrombocytopenia | interventions — Busulfan; Cyclophosphamide; fludarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (busulfan, fludarabine, HSCT, cyclophosphamide) (Experimental): Participants receive busulfan IV over 2 hours and fludarabine IV over 30 minutes on days -5 to -2. Participants undergo HSCT on day 0. Participants then receive cyclophosphamide IV over 60 minutes on days 3 and 4.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Hematopoietic Cell Transplantation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Hematopoietic Cell Transplantation — Undergo HSCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well busulfan, fludarabine, donor stem cell transplant, and cyclophosphamide in treating participants with multiple myeloma or myelofibrosis. Drugs used in chemotherapy, such as busulfan, fludarabine, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the participant they may help the participant's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving busulfan and fludarabine before and cyclophosphamide after donor stem cell may work better in treating participants with multiple myeloma or myelofibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate non-relapse mortality (NRM) up to day +100.

SECONDARY OBJECTIVES:

I. To evaluate non-relapse mortality (NRM) up to day +365. II. To evaluate the incidence of acute graft versus host disease (GVHD) and chronic GVHD up to day +365 post-transplant.

III. To evaluate the overall survival and disease free survival up to 1 year. IV. To evaluate clinical response and molecular response (complete response and partial response) up to 1 year.

OUTLINE:

Participants receive busulfan intravenously (IV) over 2 hours and fludarabine IV over 30 minutes on days -5 to -2. Participants undergo hematopoietic cell transplantation (HSCT) on day 0. Participants then receive cyclophosphamide IV over 60 minutes on days 3 and 4.

After completion of study treatment, participants are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Participants must have one of the following diagnoses of multiple myeloma (MM) or primary/secondary myelofibrosis (MF)
* Participants must have histologically documented multiple myeloma (MM)

  * Participants in early relapse (less than 24 months from initiation of systemic anti-myeloma therapy which may include single or planned tandem autologous transplant) after primary therapy that included and autologous HSCT; OR
  * Later stage; OR
  * High risk factors defined by the presence of any one of the following detected at any time prior to enrollment: deletion of chromosome 13 by conventional cytogenetics, hypodiploidy, abnormality in chromosome 1 (1q amplification or 1p deletion), t(4;14), t(14;16), t(14;20) or deletion of 17p by fluorescence in situ hybridization (FISH) or conventional karyotyping; high risk criteria based on commercially available gene expression profiling; OR
  * Extramedullary disease, plasma cell leukemia or high lactate dehydrogenase (LDH)
* Participants must have histologically documented myelofibrosis (MF)

  * Participants with Dynamic International Prognostic Scoring System (DIPSS) plus intermediate stage 2 or higher risk MF; OR
  * Subset of intermediate stage 1 participants; defined by:

    * Poor-risk molecular profile (triple negative: JAK2, CALR, MPL); OR
    * Presence of any of the following mutations: ASXL1, SRSF2, EZH2, IDH1/2; OR
    * Severe thrombocytopenia, severe anemia, high peripheral blood blasts percentage; OR
    * Unfavorable cytogenetic abnormalities (rearrangements of chromosome 5 or 7 or >= 3 abnormalities
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines
* DONOR: A related donor - fully matched
* DONOR: A related donor - haploidentical
* DONOR: An unrelated donor - fully matched
* DONOR: An unrelated donor -9/10 matched

Exclusion Criteria:

* Cardiac-left ventricular ejection fraction < 40%, symptomatic coronary artery disease, or uncontrolled arrhythmias
* Pulmonary-forced expiratory volume at one second (FEV1) or diffusion capacity of lung for carbon dioxide (DLCO) < 40% or history of chronic use of supplemental oxygen. Temporary use of supplemental oxygen at the time of screening or registration is allowed if the investigator feels that the underlying cause of requiring oxygen is reversible by the time treatment begins.
* Renal-calculated or measured glomerular filtration rate (GFR) < 30 ml/min, dialysis-dependent, or history of renal transplant
* Hepatic-bilirubin > 2 X upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 2.5 X ULN or cirrhosis
* Participants with active or uncontrolled bacterial, viral, or fungal infections requiring systemic therapy
* Pregnant women, nursing mothers or women of child-bearing potential who are unwilling to use medically accepted methods of contraception
* Male and female subjects not willing to agree to medically accepted methods of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lee, MD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Particpants - Treatment: Participants receive busulfan IV over 2 hours and fludarabine IV over 30 minutes on days -5 to -2. Participants undergo hematopoietic stem cell transplant (HSCT) on day 0. Participants then receive cyclophosphamide IV over 60 minutes on days 3 and 4.
Period: Overall Study
Arm/Group | All Particpants - Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants - Treatment: Participants receive busulfan IV over 2 hours and fludarabine IV over 30 minutes on days -5 to -2. Participants undergo hematopoietic stem cell transplant (HSCT) on day 0. Participants then receive cyclophosphamide IV over 60 minutes on days 3 and 4.
Arm/Group | All Participants - Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.17 (6.97)
Age, Continuous [Median (Full Range); unit: years] | 54.5 [50 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Non-relapse Mortality (NRM) at Day 100
Description: NRM is defined as death due to GVHD, infections, sepsis, organ (lung, liver, kidney) toxicity. Death from underlying disease (i.e. progression or relapse) is not considered NRM.
Time Frame: Up to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants - Treatment
Number analyzed (Participants) | 6
Participants | 1

2. Secondary Outcome: Non-relapse Mortality (NRM) at Day 365
Description: as for outcome 1
Time Frame: Up to day 365
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants - Treatment
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Incidence of Acute Graft Versus Host Disease (GVHD)
Description: Cases of acute graft versus host disease (GVHD) will be diagnosed by the treating physician and will be reported as a count of participants with acute GVHD.
Time Frame: Up to day 365
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 6
Participants | 2

4. Secondary Outcome: Incidence of Chronic GVHD
Description: Chronic GVHD will be assessed based on criteria established by the National Institutes of Health Consensus Development Project in 2005, and recently updated in 2014. This will be reported as a count of participants diagnosed with chronic GVHD
Time Frame: Up to day 365
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 6
Participants | 1

5. Secondary Outcome: Overall Survival at One Year
Description: Overall survival is defined as the number of participants remaining alive up to one year following stem cell transplant.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 6
Participants | 3

6. Secondary Outcome: Disease Free Survival at One Year
Description: Disease free survival is defined as an absence of disease relapse or progression up to one year following stem cell transplant.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 6
Participants | 3

7. Secondary Outcome: Number of Participants With Different Clinical Responses
Description: Clinical Responses were determined by disease-specific criteria taking into account multiple clinical and molecular markers. Multiple Myeloma (MM) response was determined using International Myeloma Working Group (IMWG) consensus criteria for response. Participants with MM had either Stringent Complete Response (sCR) or Very Good Partial Response (VGPR). Myelofibrosis (MF) response was determined using International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus criteria. Participants with MF had either Complete Response (CR) or Stable Disease (SD) (also referred to in the protocol as no response).
Time Frame: Up to 1 year
Population: one participant was not evaluable due to failure to engraft (no response assessments performed)
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 5
Participants
  Stringent Complete Response (sCR) | 1
  Very Good Partial Response (VGPR) | 1
  Complete Response (CR) | 2
  Stable Disease (SD) | 1

8. Secondary Outcome: Number of Participants With Minimal Residual Disease (MRD) Response
Description: After bone marrow transplant, bone marrow was collected every 3-6 months (as clinically indicated per treating investigator) for up to one year after bone marrow transplant. Bone marrow was evaluated by a clinical pathologist for any evidence of multiple myeloma (MM) or myelofibrosis (MF). Evidence of MM or MF in the bone marrow is referred to as minimal residual disease (MRD). A participant with evidence of MRD is MRD-positive. A participant with no evidence of MRD is MRD-negative, which is considered an MRD response. This outcome reports the number participants with MRD responses any time between bone marrow transplant up to one year of follow-up.
Time Frame: Up to 1 year
Population: one participant was not evaluable due to failure to engraft (no response assessments performed)
Measure: Count of Participants; unit: Participants
Arm/Group | All Particpants - Treatment
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected from Day -6 (6 days prior to stem cell transplant) to day +365 (365 days after stem cell transplant), approximately one year total.
Description: The occurrence of AEs was sought by non-directive questioning of the participant at each visit or phone contact, or when they were volunteered by the participant during or between visits, or through physical examination, laboratory test, or other assessments. Only G3-4 non-hematologic toxicities related to study treatment, engraftment failure, and SAEs were recorded and reported here. Relapse of disease or chronic or acute GVHD were not treated as AEs unless leading to a fatal outcome.
Arm/Group | All Participants - Treatment
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 4/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants - Treatment (N=6)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 — Engraftment Failure
Death NOS (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1 (2)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 — Sinusoidal Obstruction Syndrome
Lung infection (Infections and infestations) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Sepsis (Infections and infestations) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants - Treatment (N=6)
Anemia (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vasovagal reaction (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT03303950/Prot_SAP_000.pdf